CLINICAL TRIAL: NCT06738420
Title: Efficacy and Tolerability of a Nutritional Supplementation With Medical Nutrition Formulations Enriched With Postbiotics for the Management of Gastrointestinal Disorders: a Pilot Trial
Brief Title: Medical Nutrition Formulations Enriched With Postbiotics for the Management of Gastrointestinal Disorders
Acronym: ABB S3/ABB C22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotek (Industry)
Collaborators: Colisée Barcelona Isabel Roig (Unknown); Grupo Colisée (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-003423-18
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Diarrhoea of Diverse Aetiology Requiring Oral Rehydration Therapy; Diarrhoea and Gastrointestinal Symptoms Secondary to Enteral Nutrition
Keywords: diarrhoea; postbiotic; adults
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ABB S3 - active (Experimental): Postbiotic ABB S3 for suspension into Nutritional supplementation with Medical Nutrition Formula for the management of gastrointestinal symptoms secondary to enteral nutrition
  Interventions: Dietary Supplement: ABB S3
- ABB S3 - Placebo (Placebo Comparator): Placebo for suspension into Nutritional supplementation with Medical Nutrition Formula for the management of gastrointestinal symptoms secondary to enteral nutrition
  Interventions: Dietary Supplement: Placebo
- ABB C22 - active (Experimental): Oral Rehydration Solution containing postbiotics ABB C22 for the management of diarrhoea signs of dehydration
  Interventions: Dietary Supplement: ABB C22
- ABB C22 - placebo (Placebo Comparator): Oral Rehydration Solution containing placebo for the management of diarrhoea signs of dehydration
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ABB S3 — Postbiotic ABB S3 for suspension into Nutritional supplementation with Medical Nutrition Formula for the management of gastrointestinal symptoms secondary to enteral nutrition
  Arms: ABB S3 - active
Dietary Supplement: ABB C22 — Oral Rehydration Solution containing postbiotics ABB C22 for the management of diarrhoea signs of dehydration
  Arms: ABB C22 - active
Dietary Supplement: Placebo — Placebo for suspension into Nutritional supplementation with Medical Nutrition Formula for the management of gastrointestinal symptoms secondary to enteral nutrition
  Arms: ABB S3 - Placebo
Dietary Supplement: Placebo — Oral Rehydration Solution containing placebo for the management of diarrhoea signs of dehydration
  Arms: ABB C22 - placebo

SUMMARY:
Efficacy and tolerability of ABB i5 prebiotic and ABB C22 postbiotics for the management of constipation and gastrointestinal well-being: a pilot trial

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of the centre

  * Diagnostic of diarrhoea: increase in daily faecal weight > 200 g (as per the Centre protocol).
  * Subjects who as per the Centre protocol require Oral rehydration therapy
  * Patients with the ability to take the study product orally

Exclusion Criteria:

* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active principle or to any of the excipients.

  * History or evidence of any medical conditions or medication used that, in the opinion of the principal investigator, could affect the safety of the subjects or interfere with the study evaluations
  * Patients in situation of last days
  * Amytriptilin and masalazine treatment (anti-depressives)
  * Laxatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Faecal calprotectin | from baseline to day 14 of supplementation
  change in faecal calprotectin levels (mg/g)
faecal lactoferrin | from baseline to day 14 of supplementation
  change in the number of participants with a positive "faecal lactoferrin" result (%)
Blood IgAs | from baseline to day 14 of supplementation
  levels of serum IgAs (mg/dL)

SECONDARY OUTCOMES:
Gastrointestinal symptoms | from baseline to day 14 of supplementation
  assessment of number of diarrhea, vomits and regurgitation events
faecal consisitency | from baseline to day 14 of supplementation
  assessed through Bristol scale (1-7 score)

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Roig, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Biomarkers data (calprotectin, lactoferrin, igA) data, Bristol scale data
Supporting Information: Study Protocol
Time Frame: According to legislation

REFERENCES:
- [Derived] Mateus Rodriguez JA, Rodriguez Sanz P, Kostandyan E, Palacios Sanchez R, Pino Roque ML, Chaves Vasquez P, Roy Millan P. Mitigating Diarrhoea-Related Inflammation in Frail Older Adults with Postbiotic-Enhanced Oral Rehydration Solution: Insights from a Randomised, Double-Blind, Placebo-Controlled Study. Geriatrics (Basel). 2025 Mar 1;10(2):34. doi: 10.3390/geriatrics10020034. PMID 40126284